CLINICAL TRIAL: NCT05740956
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10502 in Patients With Advanced Solid Tumors
Brief Title: A Study of Hansoh (HS)-10502 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10502-101
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Breast Cancer; Pancreatic Cancer; Prostatic Cancer; Colorectal Cancer
Keywords: Poly(ADP-ribose) polymerase-1 inhibitor; HS-10502; Ovarian Cancer; Breast Cancer; Prostate Cancer, Colorectal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10502 (Experimental): HS-10502 Tablets，PO，QD
  Interventions: Drug: HS-10502

INTERVENTIONS:
Drug: HS-10502 — HS-10502 will be administered once per day on a continuous dosing schedule starting on Cycle 1 Day 1 (C1D1) in a 28-day treatment cycle.

SUMMARY:
HS-10502 is a Poly(ADP-ribose) polymerase 1 (PARP1)-specific selective inhibitor. The purpose if this study is to assess the safety, tolerability, pharmacokinetics (PK), and efficacy of HS-10502 in subjects with homologous recombination repair (HRR) gene mutant or homologous recombination deficiency (HRD) positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 - 75 years (inclusive).
2. Having at least one target lesion per the RECIST v1.1.
3. For the phase Ia Cohort A: advanced solid tumor carrying HRR gene mutation with failure or intolerance or not available to the currently available Standard of care (SoC).
4. For the phase Ib study:

   Cohort B: patients with HRD positive recurrent ovarian cancer with failure or intolerance or not available to SoC Cohort C: patients with HRR gene mutation advanced Human epidermal growth factor receptor 2 (HER2)-negative breast cancer with failure or intolerance or not available to SoC Cohort D: patients with HRR gene mutation advanced pancreatic cancer with failure or intolerance or not available to SoC Cohort E: patients with HRR gene mutation mCRPC with failure or intolerance or not available to SoC Cohort F: patients with HRR gene mutation colorectal cancer with failure or intolerance or not available to SoC Cohort G: patients with other HRR gene mutation or HRD positive advanced solid tumors with failure or intolerance or not available to SoC
5. Eastern cooperative oncology group (ECOG) performance status was 0-1.
6. Minimum life expectancy > 12 weeks.
7. Females should be using adequate contraceptive measures and should not be breastfeeding Males should be using adequate contraceptive measures.
8. Have signed Informed Consent Form.

Exclusion Criteria:

1. Received or are receiving the following treatments:

   1. Previous or current treatment with two or more Poly(ADP-ribose) polymerase (PARP) inhibitors.
   2. Traditional Chinese medicine indicated for tumors within 2 weeks prior to the first dose of study treatment.
   3. Cytotoxic chemotherapeutic drugs, investigational drugs or other systematic anti-tumor therapies within 3 weeks before the first dose of study treatment; Nitrosourea or Mitomycin C within 6 weeks prior to the first dose of study treatment.
   4. Local radiotherapy within 2 weeks prior to the first dose of study treatment; more than 30% of bone marrow radiotherapy or large-area irradiation within 4 weeks before the first dose of study treatment.
   5. Presence of pleural effusion/ascites requiring clinical intervention; presence of pericardial effusion.
   6. Major surgery within 4 weeks prior to the first dose of study treatment.
2. Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
3. History of other primary malignancies.
4. Known and untreated, or active central nervous system metastases.
5. Inadequate bone marrow reserve or hepatic and renal functions.
6. Myelodysplastic syndromes (MDS) or acute myeloid leukemia (AML), or with features suggestive of MDS or AML.
7. Severe, uncontrolled or active cardiovascular disorders.
8. Diabetic ketoacidosis or hyperosmolar hyperglycemic state within 6 months prior to the first dose of study treatment; glycosylated hemoglobin ≥ 7.5%.
9. Serious or poorly controlled hypertension.
10. Any life-threatening hemorrhagic event or events requiring blood transfusion within 120 days prior to the first dose of study treatment. Clinically significant hemorrhagic symptoms or obvious hemorrhagic tendency.
11. Serious infection within 4 weeks prior to the first dose of study treatment, or presence of uncontrollable active infection in the screening period.
12. Having serious neurological or mental disorders.
13. A history of hypersensitivity to any of the active or inactive ingredients of HS-10502 or drugs with a similar chemical structure to HS-10502 or in the same class as HS-10502.
14. Patients who may have poor compliance with the procedures and requirements of the study, as judged by the investigator.
15. Patients with any condition that jeopardizes the safety of the patient or interferes with the assessment of the study, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HS-10502（Stage 1） | Cycle 1 (28 days)
  MTD is defined as the previous dose level at which 2 or more out of 2-6 subjects experienced a Dose-limiting toxicity (DLT)
Maximum applicable dose (MAD) of HS-10502（Stage 1） | Cycle 1 (28 days)
  MAD is defined as follows: a) based on PK data, it is anticipated that at this dose level, the dose-exposure plateau has been reached, b) based on existing safety data, it is judged that dose escalation following this dose level will have a large safety risk or subject intolerance, or c) based on the pharmacokinetics-pharmacodynamics (PK-PD) model, it suggested that the optimal target concentration of safety and efficacy has been explored
Efficacy of HS-10502: Objective response rate (ORR)（Stage 2） | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  ORR is defined as the proportion of participants with Best Overall Response (BOR) of confirmed CR or confirmed PR per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only)

SECONDARY OUTCOMES:
[Stage 1 and Stage 2] Incidence and severity of treatment-emergent adverse events | From Cycle 1 Day 1 (C1D1) until 28 days after the final dose. A cycle is 28 days
  Assessed by number and severity of adverse events as evaluated according to NCI CTCAE v5.0.
[Stage 1 and Stage 2] PK parameters: The maximum observed concentration (Cmax) of HS-10502 | Cycle 1 Day 1 (each cycle is 28 days)
  Maximum plasma drug concentration of HS-10502
[Stage 1 and Stage 2] PK parameters: time to Cmax (Tmax) of HS-10502 | Cycle 1 Day 1 (each cycle is 28 days)
  Time of maximum observed concentration of HS-10502
[Stage 1 and Stage 2] PK parameters: area under the concentration-time curve from time 0 to time t of last measurable concentration (AUC0-t) of HS-10502 | Cycle 1 Day 1 (each cycle is 28 days)
  Area under the curve from the time of dosing to the time of the last measurable (positive) concentration
[Stage 1 and Stage 2] PK parameters: Maximum plasma concentration at steady state (Css, max) of HS-10502 | Cycle 2 Day 1 (each cycle is 28 days)
  Maximum plasma drug concentration at steady state of HS-10502.
[Stage 1 and Stage 2] PK parameters: time to Css, max (Tss, max) of HS-10502 | Cycle 2 Day 1 (each cycle is 28 days)
  Time of maximum observed concentration at steady state of HS-10502
[Stage 1 and Stage 2] PK parameters: Minimum plasma concentration at steady state (Css, min) of HS-10502 | Cycle 2 Day 1 (each cycle is 28 days)
  Minimum plasma drug concentration at steady state of HS-10502
[Stage 1 and Stage 2] PK parameters: Area under the plasma concentration-time curve over a dosing interval at steady state (AUCss) of HS-10502 | Cycle 2 Day 1 (each cycle is 28 days)
  The partial area from dosing time to dosing time plus dosing interval of HS-10502
Efficacy of HS-10502: ORR | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  Proportion of participants with BOR of confirmed CR or confirmed Partial Response (PR) per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and The prostate cancer working group 3 criteria (PCWG3) (for prostate cancer only)
[Stage 1 and Stage 2] Efficacy of HS-10502: disease control rate (DCR) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  P Percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks) per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only)
Title: [Stage 1 and Stage 2] Efficacy of HS-10502: duration of response (DoR) | From the date of CR, PR until the date of disease progression or withdrawal from study, approximately 2 years
  DoR only applies to participants whose best overall response is CR or PR based on assessment per RECIST v1.1 (applicable for all solid tumors except prostate cancer) or per RECIST v1.1 and PCWG3 (for prostate cancer only). The start date is the date of first documented response of CR or PR (i.e. the start date of observed response, not the date when response was confirmed), and the end date is the date of the first documented progression or death due to underlying cancer.
[Stage 1 and Stage 2] Efficacy of HS-10502: progression free survival (PFS) (applicable for all solid tumors except prostate cancer) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or withdrawal from study, approximately 2 years.
  Time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. PFS will be assessed per RECIST v1.1.
[Stage 1 and Stage 2] Efficacy of HS-10502: radiographic progression free survival (rPFS) (for prostate cancer only) | From the date of randomization or first dose (if randomization is not needed) until the date of disease progression or withdrawal from study, approximately 2 years
  Time from the date of randomization or first dose (if randomization is not needed) to the date of the first documented progression or death due to any cause. rPFS will be assessed per RECIST v1.1 (soft tissue) and PCWG3 (bone).
[Stage 1 and Stage 2] Efficacy of HS-10502: ORR evaluated by RECIST v1.1 and Gynecologic Cancer Intergroup (GCIG) CA-125 (for ovarian cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  Proportion of participants with BOR of confirmed CR or confirmed PR per both RECIST v1.1 and GCIG CA-125 criteria.
[Stage 2] Efficacy of HS-10502: overall survival (OS) | From the date of randomization or first dose (if randomization is not needed) until the documentation of death from any cause, approximately 4 years
  Time from the date of randomization or first dose (if randomization is not needed) to the date of death due to any cause. For each participant who is not known to have died as of the cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive
[Stage 1 and Stage 2] Efficacy of HS-10502: Proportion of subjects with Carbohydrate antigen (CA)-125 decreased by ≥ 50% from baseline (for ovarian cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  The percentage of subjects (ovarian cancer only) with a reduction of at least 50% from baseline in CA-125 levels.
[Stage 1 and Stage 2] Efficacy of HS-10502: ≥ 50% PSA decrease (PSA50) response rate (for prostate cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  Proportion of subjects with a Prostate-specific antigen (PSA) nadir of ≤ 50% of baseline PSA level confirmed by serial PSA assessments (at least 3 weeks apart) after the start of the study.
[Stage 1 and Stage 2] Efficacy of HS-10502: Time to PSA progression (for prostate cancer only) | From the date of first dose until the date of disease progression or withdrawal from study, approximately 2 years
  Time from the first dose to PSA progression based on PCWG3 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Acedemy of Medical Sciences, Beijing, Beijing Municipality, China